CLINICAL TRIAL: NCT04026789
Title: Medication Abortion for Pregnancy of Unknown Location
Acronym: MAPUL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000848
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (plus prospective cohort for those interested in participation but unwilling to be randomized)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same-day-start (Active Comparator): Patients seeking medication abortion who are shown to have an asymptomatic, low-risk pregnancy of unknown location who are randomized to same-day start will have their medication abortion initiated on the day that they present for services while simultaneously ruling out ectopic pregnancy with serial hcg testing
  Interventions: Other: Same-day-start
- Delay-for-diagnosis (Active Comparator): Patients seeking medication abortion who are shown to have an asymptomatic, low-risk pregnancy of unknown location who are randomized to delay-for-diagnosis will first have ectopic pregnancy ruled out with serial hcg and ultrasounds prior to initiating medication abortion
  Interventions: Other: Delay-for-diagnosis

INTERVENTIONS:
Other: Same-day-start — Patients seeking medication abortion who are shown to have an asymptomatic, low-risk pregnancy of unknown location who are randomized to same-day start will have their medication abortion initiated on the day that they present for services while simultaneously ruling out ectopic pregnancy with serial hcg testing
  Arms: Same-day-start
Other: Delay-for-diagnosis — Patients seeking medication abortion who are shown to have an asymptomatic, low-risk pregnancy of unknown location who are randomized to delay-for-diagnosis will first have ectopic pregnancy ruled out with serial hcg and ultrasounds prior to initiating medication abortion
  Arms: Delay-for-diagnosis

SUMMARY:
The purpose of this study is to compare time to completed abortion between two protocols for patients seeking medication abortion - same-day start versus delay-for-diagnosis - in the setting of asymptomatic, low-risk, pregnancy of unknown location.

ELIGIBILITY:
Patients with an undesired pregnancy of less than or equal to 42 days gestation based on last menstrual period (LMP) who present to Planned Parenthood League of Massachusetts (PPLM)'s Greater Boston Health Center seeking medication abortion will be considered for study participation.

Inclusion criteria:

* Positive urine or serum hCG test
* No evidence of gestational sac on transvaginal ultrasound
* Desire for medication abortion as method of pregnancy termination

Exclusion criteria:

* Ineligible for medication abortion at PPLM based on current PPLM clinical guidelines
* Reasonable clinical suspicion for ectopic or molar pregnancy, such as abnormal or concerning ultrasound findings
* High risk for ectopic pregnancy, such as prior ectopic pregnancy, history of tubal surgery, concurrent intrauterine device in place during this pregnancy
* Exhibiting symptoms of possible ectopic, such as vaginal bleeding or abdominal pain
* LMP > 42 days or unknown LMP
* Age less than 18 years
* Prior participation in this study
* Anticipated inability to present for scheduled follow-up visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-07-17 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to completed abortion | through study completion, an average of two weeks
  Time to completed abortion as defined by the number of days between initial ultrasound diagnosis of PUL to the diagnostic test that confirms complete abortion

SECONDARY OUTCOMES:
Number of participants with complete expulsion of pregnancy without surgical intervention | 14 days after initiation of medical abortion
  Efficacy of medical abortion, defined as number of participants with complete expulsion of pregnancy without surgical intervention
Time to diagnosis of pregnancy outcome | Within 2 weeks of identification of pregnancy of unknown location on ultrasound
  Number of days between initial ultrasound diagnosis of pregnancy of unknown location and diagnosis of pregnancy outcome, with options including intrauterine pregnancy, ectopic pregnancy, or early pregnancy loss
Rate of ectopic pregnancy | Within 2 weeks of identification of pregnancy of unknown location on ultrasound
  Rate of ectopic pregnancy among entire study population
Percent of participants who complete follow-up and confirm complete abortion | Within 1 month of identification of pregnancy of unknown location on ultrasound
  Percent of participants who adhered to recommended follow-up plan and confirmed a complete abortion through ultrasound or hCG

CONTACTS AND LOCATIONS:
Locations (1):
- PPLM, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with any other researchers.